CLINICAL TRIAL: NCT01640301
Title: Phase I/II Study of Adoptive Immunotherapy After Allogeneic HCT With Virus Specific CD8+ T Cells That Have Been Transduced to Express a WT1-Specific T Cell Receptor for Patients With Relapsed AML
Brief Title: Laboratory-Treated T Cells in Treating Patients With High-Risk Relapsed Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Chronic Myelogenous Leukemia Previously Treated With Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Associate Professor, Program in Immunology, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2498.00; NCI-2011-03362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2498; 2498.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); RG9212029 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2011-11-29; First posted 2012-07-13 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia; Donor; Hematopoietic Cell Transplant Recipient; HLA-A*0201 Positive Cells Present; Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (high-risk for relapse after HCT) (Experimental): Patients with no evidence of leukemia or MDS post-HCT receive WT1-sensitized T cells IV over 45 minutes (or longer for patients who are 15-30 kg) on days 0 and 14 and aldesleukin SC BID on days 14-28.
  Interventions: Biological: Aldesleukin; Other: Laboratory Biomarker Analysis; Biological: WT1-Sensitized Allogeneic T-Lymphocytes
- Arm II (relapsed after HCT) (Experimental): Patients with evidence of AML (minimal residual disease or overt relapse) post-HCT receive cyclophosphamide IV and fludarabine phosphate IV daily on days -4 to -2. Patients also receive WT1-sensitized T cells IV over 45 minutes (or longer for patients who are 15-30 kg) on days 0 and 21 and aldesleukin SC BID on days 14-28.
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: WT1-Sensitized Allogeneic T-Lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm II (relapsed after HCT)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
  Arms: Arm II (relapsed after HCT)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: WT1-Sensitized Allogeneic T-Lymphocytes — Given IV

SUMMARY:
This phase I/II trial studies the side effects of laboratory-treated T cells and to see how well they work in treating patients with high-risk acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelogenous leukemia (CML) that has returned after a period of improvement (relapsed), previously treated with donor stem cell transplant. Biological therapies, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop cancer cells from growing. Placing a gene that has been created in the laboratory into a person's T cells may make the body build an immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and potential toxicities associated with treating patients with high risk or relapsed AML, MDS, and CML after allogeneic hematopoietic cell transplantation (HCT) by adoptive transfer of virus-specific cluster of differentiation (CD)8 T cells genetically-modified to express a high affinity Wilms tumor 1 (WT1)-specific T cell receptor (TCR).

II. Determine the anti-leukemic activity associated with treating patients with relapsed AML, MDS and CML after allogeneic HCT by adoptive transfer of virus-specific CD8 T cells genetically-modified to express a high affinity WT1-specific T cell receptor (TCR).

SECONDARY OBJECTIVES:

I. Determine the in vivo persistence of transferred T cells and ability to migrate to and accumulate in bone marrow.

II. Determine the maintenance of TCR expression and function of transduced T cells.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients with no evidence of leukemia post-HCT receive WT1-sensitized T cells intravenously (IV) over 45 minutes (or longer for patients who are 15-30 kg) on days 0 and 14 and aldesleukin subcutaneously (SC) twice daily (BID) on days 14-28.

ARM II: Patients with evidence of AML (minimal residual disease or overt relapse) post-HCT receive cyclophosphamide IV and fludarabine phosphate IV daily on days -4 to -2. Patients also receive WT1-sensitized T cells IV over 45 minutes (or longer for patients who are 15-30 kg) on days 0 and 21 and aldesleukin SC BID on days 14-28.

After completion of study treatment, patients are followed up weekly for 4 weeks, at weeks 6 and 8, at 3, 6, 12 months, and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must express HLA-A*0201
* Patients who are currently undergoing or who previously underwent matched allogeneic HCT for:

  * AML: Prospective enrollment will now be limited to patients with relapsed disease (overt relapse or minimal residual disease) at any time post allogeneic HCT
  * MDS will no longer be a criterion for eligibility
  * CML will no longer be a criterion for eligibility
* Patients must have an HLA-matched donor of hematopoietic stem cells (related or unrelated)
* Patients must be able to provide blood and bone marrow samples and undergo the procedures required for this protocol
* Patients must be >= 15 kg, as patients with lower weight would be incapable of providing high volume and frequent blood samples for monitoring and analysis
* Patients must be able to give informed consent; parent or legal representative will be asked to consent for patients younger than 18 year old
* DONOR: Patient and donor (related or unrelated) must be HLA-matched and express HLA-A*0201
* DONOR: Donor must be Epstein-Barr virus (EBV) or cytomegalovirus (CMV) seropositive
* DONOR: Donor must be age 18 or older
* DONOR: In good general health
* DONOR: Able to give informed consent

Exclusion Criteria:

* Central nervous system (CNS) tumor refractory to intrathecal chemotherapy and/or cranio-spinal radiation
* In patients whose leukemic cells are available for evaluation, the expression of WT1 in the patient's bone marrow will be determined; if WT1 expression in the patient's bone marrow is not highly expressed by polymerase chain reaction (PCR), the patient will be excluded from the study; patients with no evaluable leukemia will be eligible for enrollment based on the high frequency of positive leukemias (> 90%), and leukemia will be evaluated for WT1 expression if recurrence is detected
* Human immunodeficiency virus (HIV) seropositive; testing for HIV should be within 6 months of enrollment
* Medical or psychological conditions that would make the patient unsuitable candidate for cell therapy at the discretion of the principal investigator (PI)
* Pregnancy or breast-feeding; women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (B-hCG) pregnancy test result within 14 days before the first dose of WT1-specific T cell infusion; woman of non-childbearing potential will be defined as being postmenopausal greater than one year or who have had a bilateral tubal ligation or hysterectomy; all recipients of WT1-specific T cells will be counseled to use effective birth control during participation in this study and for 12 months after the last T cell infusion
* DONOR: Less than 18 years old
* DONOR: Active infectious hepatitis
* DONOR: HIV or human T-lymphotropic virus (HTLV) seropositive
* DONOR: Pregnancy or nursing
* DONOR: Significant medical conditions (e.g. immunosuppressive therapy) that would make the donor an unsuitable T cell donor
* DONOR: Unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chapuis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Chapuis AG, Egan DN, Bar M, Schmitt TM, McAfee MS, Paulson KG, Voillet V, Gottardo R, Ragnarsson GB, Bleakley M, Yeung CC, Muhlhauser P, Nguyen HN, Kropp LA, Castelli L, Wagener F, Hunter D, Lindberg M, Cohen K, Seese A, McElrath MJ, Duerkopp N, Gooley TA, Greenberg PD. T cell receptor gene therapy targeting WT1 prevents acute myeloid leukemia relapse post-transplant. Nat Med. 2019 Jul;25(7):1064-1072. doi: 10.1038/s41591-019-0472-9. Epub 2019 Jun 24. PMID 31235963
- [Derived] Oda SK, Daman AW, Garcia NM, Wagener F, Schmitt TM, Tan X, Chapuis AG, Greenberg PD. A CD200R-CD28 fusion protein appropriates an inhibitory signal to enhance T-cell function and therapy of murine leukemia. Blood. 2017 Nov 30;130(22):2410-2419. doi: 10.1182/blood-2017-04-777052. Epub 2017 Oct 17. PMID 29042364

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 participants were enrolled on the study, meaning they signed the consent for treatment. However, 19 did not move on to treatment for various reasons.
Period: Overall Study
Arm/Group | Arm I (High-risk for Relapse After HCT) | Arm II (Relapsed After HCT)
Started | 13 | 15
Completed | 13 | 7
Not Completed | 0 | 8
Not completed — Death | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (High-risk for Relapse After HCT) | Arm II (Relapsed After HCT) | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Anti-leukemic Potential Efficacy, in Terms of Duration of Response (Arm II)
Description: Response is assessed throughout the 1 year post treatment timeframe. Morphologic criteria for response:
  Complete Response (CR) = Bone Marrow blasts <5%; no blasts with Auer rods; no extramedullary disease. Transfusion independent.
  Platelets ≥ 100,000/μl Absolute neutrophil count >1000/μl (CRi: incomplete hematologic recovery CRp: incomplete platelet recovery)
  Partial Response (PR) = Decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow and the normalization of blood counts as for CR. (PRi and PRp if incomplete hematologic or platelet recovery)
  Stable Disease (SD) = Failure to achieve at least PR, but no evidence of progression for >4 weeks.
Time Frame: Up to 1 year
Population: 4 patients in Arm II did not relapse and were not assessed. 1 pt progressed at their D365 visit timepoint which landed on D367. They were included in the count of participants that passed within their 1 year follow-up timeframe.
Measure: Median (Full Range); unit: days
Groups:
- Group 2 (Avelumab, MHC Class I Up-regulation, T Cells): Patients who have an HLA type for which T cells can be generated receive avelumab IV over 1 hour every 2 weeks for 12 months. Patients also receive MHC class I up-regulation intervention as in Group 1 between 7-10 days after the first infusion of avelumab and 2-5 days before the first infusion of MCPyV TAg-specific polyclonal autologous CD8+ T cells. Patients receive two infusions of MCPyV TAg-specific polyclonal autologous CD8+ T cells IV over 60-120 minutes.
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 9
days | 28 [5 to 367]

2. Primary Outcome: Efficacy, in Terms of Relapse Rate (Arm I)
Time Frame: At 1 year post-transplant
Population: No patients in Arm I relapsed, so overall number of participants analyzed is 0
Groups:
- Group 1 (Avelumab and MHC Class I Up-regulation): Patients who do not have a HLA type for which T cells can be generated or for whom T cells cannot be generated for technical issues receive avelumab intravenously (IV) over 1 hour every 2 weeks for 12 months. Within 7-10 days after completion of 1-3 doses of avelumab, patients receive MHC class I up-regulation intervention comprising either localized radiation therapy or recombinant interferon beta via intra-tumor injection.
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 0

3. Primary Outcome: Count of Participants Who Experienced Chronic Graft Versus Host Disease (GVHD) (Arm I)
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 12
Participants | 6

4. Primary Outcome: Count of Participants Who Experienced Chronic Graft Versus Host Disease (GVHD) (Arm II)
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 15
Participants | 8

5. Primary Outcome: Count of Participants Who Experienced Grade III-IV Acute Graft Versus Host Disease (GVHD) (Arm II)
Time Frame: Up to 1 year following infusion per patient
Population: 2 patients were unevaluable for this outcome due to old documentation, unable to discern if the patient had acute GvHD greater than or equal to grade 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 13
Participants | 0

6. Primary Outcome: Count of Participants Who Experienced Grade III-IV Acute Graft-versus-host Disease (GVHD) (Arm I)
Time Frame: Up to 1 year
Population: All patients were evaluated for aGvHD greater than or equal to Grade 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 13
Participants | 1

7. Primary Outcome: Treatment-related Toxicity Rate (Arm I)
Description: Outcome will be reported as a count of participants that experienced adverse events. Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Time Frame: Up to 30 days after last study intervention per patient
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 13
Participants | 12

8. Primary Outcome: Treatment-related Toxicity Rate (Arm II)
Description: as for outcome 7
Time Frame: Up to 30 days after last study intervention per patient
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 15
Participants | 15

9. Secondary Outcome: Disease-free Survival After T Cell Therapy
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (High-risk for Relapse After HCT) | Arm II (Relapsed After HCT)
Number analyzed (Participants) | 13 | 15
Participants | 13 | 7

10. Secondary Outcome: Incidence of Relapse After T Cell Therapy (Arm II)
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 15
Participants | 9

11. Secondary Outcome: Maintenance of T Cell Receptor (TCR) Expression of Transduced T Cells (Arm I) i.e. Persistence
Time Frame: Up to 28 days post intervention per patient
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 12
Participants | 12

12. Secondary Outcome: Maintenance of Function of Transduced T Cells (Arm I)
Time Frame: Up to 28 days post intervention per patient
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 12
Participants | 9

13. Secondary Outcome: Time to Progression After T Cell Therapy (Arm I)
Time Frame: Up to 1 year
Population: No patients analyzed because no patients relapsed in Arm I
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year post infusion per patient
Description: Toxicities were according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.
Arm/Group | Arm I (High-risk for Relapse After HCT) | Arm II (Relapsed After HCT)
All-Cause Mortality (participants affected / at risk) | 0/13 | 8/15
Serious Adverse Events (participants affected / at risk) | 5/13 | 5/15
Other Adverse Events (participants affected / at risk) | 12/13 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (High-risk for Relapse After HCT) (N=13) | Arm II (Relapsed After HCT) (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
CPK Increased (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Sclerosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (High-risk for Relapse After HCT) (N=13) | Arm II (Relapsed After HCT) (N=15)
Anemia (Blood and lymphatic system disorders) | 4 (16) | 8 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 | 2 (2)
Nausea (Gastrointestinal disorders) | 0 | 2 (2)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (2) | 0 (0)
CANDIDA KRUSEI (Infections and infestations) | 0 | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (13) | 8 (15)
Neutrophil count decreased (Investigations) | 2 (2) | 12 (20)
Platelet count decreased (Investigations) | 2 (2) | 12 (20)
White blood cell decreased (Investigations) | 0 | 8 (13)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (5) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Hypertension (Vascular disorders) | 3 (5) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT01640301/Prot_SAP_000.pdf